CLINICAL TRIAL: NCT01859832
Title: Validation of a Novel Diagnostic Tool for the Evaluation of Post Renal Transplant Immunosuppression: The ImmuKnow Assay
Status: Completed | Type: Observational
Sponsor: London Health Sciences Centre Research Institute OR Lawson Research Institute of St. Joseph's (Other)
Collaborators: Astellas Pharma Canada, Inc. (Industry)
Responsible Party: Principal Investigator, Patrick Luke, Dr. Patrick Luke, MD, London Health Sciences Centre Research Institute OR Lawson Research Institute of St. Joseph's
Other Study IDs: R-09-016; 15785E (Other: REB)
Record Dates: First submitted 2012-05-02; First posted 2013-05-22 (Estimated); Last update posted 2015-09-02 (Estimated); Status verified 2015-08

CONDITIONS: Renal Transplant Recipients
Keywords: renal transplant; kidney transplantation; immune status; immunosuppressive medications

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Biospecimen Retention: None Retained — Collected blood samples will be discarded immediately following testing
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- Enrolled participants: All participants enrolled in this study will have been previously consented to the study entitled, "A Comparison of Effects of Standard Dose vs Low Dose Advagraf with Il-2 Receptor Antibody Induction, MMF and Steroids, With or Without ACEi/ARB-based Antihypertensive Therapy on Renal Allograft Histology, Function, and Immune Response." This is an observational study with only one group/cohort in which all participants have bloodwork collected pre-transplant and at various time points post-transplant and these samples are analyzed using the Cylex ImmuKnow Assay.
  Interventions: Other: Cylex ImmuKnow Assay

INTERVENTIONS:
Other: Cylex ImmuKnow Assay — This is not an interventional study. However the assay being tested on the samples of all enrolled participants in the Cylex ImmuKnow Assay

SUMMARY:
Patients undergoing renal transplantation at London Health Sciences Centre, University Hospital and who are participating in the study "A Comparison of Effects of Standard Dose vs Low Dose Advagraf with IL-2 Receptor Antibody Induction, MMF and Steroids, With or Without ACEi/ARB-based Antihypertensive Therapy on Renal Allograft Histology, Function, and Immune Response" will be evaluated with the ImmuKnow Assay to assess the ability of this assay to predict underimmunosuppression (rejection) or overimmunosuppression determined by this test and to determine retrospectively whether decision making utilizing this novel assay would have improved outcomes over standard techniques.

This study is designed to evaluate an in vitro assay (Cylex®ImmuKnow Assay) for the measurement of cell-mediated immune response in renal transplant patients receiving immunosuppressive therapy. This assay measures ATP as an activation response of CD4+ cells to stimulation with phytohemagglutinin (PHA) in whole blood samples as a reflection of the immune system of the patient at any point in therapy. The natural history of the immune status of the renal transplant recipient as reflected by the ImmuKnow assay will be determined at specific time points of interest including: pre and post transplant, as an adjunct to therapeutic drug monitoring, and pre and post infectious or rejection episode. Analysis of the results of the assay at these time points will allow us to retrospectively study the effects of routine immunosuppressive agent modulation on immune function, and its subsequent effects in times of renal allograft insult.

ELIGIBILITY:
Inclusion Criteria:

* Patients undergoing implantation surgery for renal transplantation at London Health Sciences Centre, University Hospital
* Patients who have consented to the study entitled, "A Comparison of Effects of Standard Dose vs Low Dose Advagraf with IL-2 Receptor Antibody Induction, MMF and Steroids, With or Without ACEi/ARB-based Antihypertensive Therapy on Renal Allograft Histology, Function, and Immune Response" Exclusion Criteria:

Exclusion Criteria:

* None

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: All participants enrolled in this study will be undergoing renal transplantation and will have already been consented to the study entitled, "A Comparison of Effects of Standard Dose vs Low Dose Advagraf with IL-2 Receptor Antibody Induction, MMF and Steroids, With or Without ACEi/ARB-based Antihypertensive Therapy on Renal Allograft Histology, Function, and Immune Response."
Sampling Method: Non-Probability Sample
Enrollment: 19 (Actual)
Dates: Start 2010-05; Primary Completion 2013-12 (Actual); Study Completion 2013-12 (Actual)

PRIMARY OUTCOMES:
Immune status | A sample will be collected pre-transplant as well as for an expected average of 6 months post-transplant.

CONTACTS AND LOCATIONS:
Overall Officials: Patrick Luke, MD, FRCSC, Principal Investigator — London Health Sciences Centre Research Institute OR Lawson Research Institute of St. Joseph's
Locations (1):
- London Health Sciences Centre, University Hospital, London, Ontario, Canada